CLINICAL TRIAL: NCT06946407
Title: A Prospective, Single-Arm Clinical Study of Rituximab, Methotrexate, and Thiotepa (R-MT) Induction Followed by Etoposide and Cytarabine (EA) Consolidation for Primary Central Nervous System Lymphoma
Brief Title: Rituximab, Methotrexate, and Tepadina Induction Followed by Etoposide and Cytarabine Consolidation in Primary Central Nervous System Lymphoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FengYan Jin (Other)
Responsible Party: Sponsor-Investigator, FengYan Jin, Clinical Professor of Hematology Department, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCNSL-RMTEA
Record Dates: First submitted 2025-04-09; First posted 2025-04-27 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Primary Central Nervous System Lymphoma (PCNSL); CNS Lymphoma Treatment
Keywords: PCNSL; Induction Therapy; Consolidation Therapy
MeSH Terms: interventions — Rituximab; Methotrexate; Thiotepa; Cytarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Evaluation of Objective Response Rate (ORR) with RMT-EA as First-Line Treatment for PCNSL (Experimental): This arm evaluates the RMT-EA regimen for first-line treatment of newly diagnosed Primary Central Nervous System Lymphoma (PCNSL).
  Pre-induction Therapy (R-M regimen):
  Cycle 1-2 (C1-C2):
  Rituximab (R): 375 mg/m² IV, on Day 1 Methotrexate (MTX): 3.5 g/m² IV over 3 hours, on Day 2
  Induction Therapy (R-MT regimen):
  Cycle 3-6 (C3-C6):
  Rituximab (R): 375 mg/m² IV, on Day 1 Methotrexate (MTX): 3.5 g/m² IV over 3 hours, on Day 2 Thiotepa (T): 30 mg/m² IV over 30 minutes, on Day 3
  Consolidation Therapy (EA regimen):
  Cycle 7-8 (C7-C8):
  Etoposide (E): 5 mg/kg IV, every 12 hours on Days 1 and 2 Cytarabine (A): 2.0 g/m² IV over 2 hours, every 12 hours on Days 3 and 4 This study arm is designed to assess the Objective Response Rate (ORR), as well as the safety, efficacy, and quality of life outcomes of the RMT-EA regimen in patients with newly diagnosed PCNSL aged ≤60 years. The dosing schedules and drug combinations outlined above distinguish this arm from others in the study.
  Interventions: Drug: Rituximab, Methotrexate, and Thiotepa (R-MT) Induction Followed by Etoposide and Cytarabine (EA) Consolidation

INTERVENTIONS:
Drug: Rituximab, Methotrexate, and Thiotepa (R-MT) Induction Followed by Etoposide and Cytarabine (EA) Consolidation — Pre-induction Therapy (R-M regimen):
  Cycle 1-2 (C1-C2):
  Rituximab (R): 375 mg/m² IV, on Day 1 Methotrexate (MTX): 3.5 g/m² IV over 3 hours, on Day 2
  Induction Therapy (R-MT regimen):
  Cycle 3-6 (C3-C6):
  Rituximab (R): 375 mg/m² IV, on Day 1 Methotrexate (MTX): 3.5 g/m² IV over 3 hours, on Day 2 Thiotepa (T): 30 mg/m² IV over 30 minutes, on Day 3
  Consolidation Therapy (EA regimen):
  Cycle 7-8 (C7-C8):
  Etoposide (E): 5 mg/kg IV, every 12 hours on Days 1 and 2 Cytarabine (A): 2.0 g/m² IV over 2 hours, every 12 hours on Days 3 and 4

SUMMARY:
High-dose methotrexate (HD-MTX) remains the foundation of treatment for primary central nervous system lymphoma (PCNSL), but outcomes are suboptimal. The addition of rituximab has shown mixed results, partly due to limited blood-brain barrier penetration. The MATRix regimen (rituximab, HD-MTX, cytarabine, thiotepa) has improved survival but is associated with significant toxicity.

Consolidation therapy is recommended after induction, but there is no standard approach. Preliminary data suggest that etoposide and cytarabine (EA) consolidation after rituximab-HD-MTX induction may offer improved tolerability, though relapse rates remain high.

This study evaluates the safety, efficacy, and tolerability of a novel RMT-EA regimen-rituximab, methotrexate, and thiotepa (RMT) induction followed by etoposide and cytarabine (EA) consolidation-in newly diagnosed, untreated PCNSL patients. The aim is to improve remission depth and prolong disease-free survival, especially in younger patients.

DETAILED DESCRIPTION:
A retrospective analysis conducted at the study center demonstrated an objective response rate (ORR) of 64.3% among patients with primary central nervous system lymphoma (PCNSL) receiving chemotherapy. This prospective, single-arm clinical study is designed to evaluate the safety, efficacy, and tolerability of a novel treatment regimen-rituximab, methotrexate, and thiotepa (RMT) for induction, followed by etoposide and cytarabine (EA) for consolidation-in patients with newly diagnosed PCNSL.

The study hypothesizes that the RMT-EA regimen will increase the ORR to 84% while maintaining an acceptable safety profile. The goal is to generate additional evidence to support the optimization of frontline therapy for PCNSL, with a focus on improving remission depth, minimizing relapse rates, and extending progression-free survival, particularly in younger patient populations.

ELIGIBILITY:
Inclusion Criteria:

* Age ≤ 60 years, male or female
* Histologically and immunohistochemically confirmed diagnosis of diffuse large B-cell lymphoma (DLBCL) without prior treatment
* No evidence of systemic lymphatic or hematopoietic involvement or other systemic disease, based on thorough physical examination and imaging/laboratory tests
* Diagnosis meets criteria for Primary Central Nervous System Lymphoma (PCNSL)
* Written informed consent obtained from the patient or their legal guardian
* Voluntary agreement to participate in the study

Exclusion Criteria:

* Presence of another active malignancy
* Known history of HIV infection or diagnosis of acquired immunodeficiency syndrome (AIDS)
* Known allergy to any of the investigational drugs or their excipients
* Any condition that, in the opinion of the investigator, may lead to early study termination, including but not limited to:
* Severe comorbidities
* Significant laboratory abnormalities
* Serious social or family circumstances affecting safety or compliance

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 41 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2029-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From the date of enrollment until the end of induction and consolidation treatment, assessed up to approximately 8 months.
  Objective Response Rate (ORR): Defined as the proportion of participants who achieve Complete Remission (CR), Unconfirmed Complete Remission (CRu), or Partial Remission (PR) according to the International Primary CNS Lymphoma Collaborative Group (IPCG) efficacy assessment criteria.

SECONDARY OUTCOMES:
Progression-Free Survival (PFS) | From the start of treatment until the first documented disease progression, treatment failure, or death, assessed up to 36 months.
  Progression-Free Survival (PFS):Defined as the time from the start of treatment to the first occurrence of disease progression, treatment failure, or death. Disease progression or failure will be defined according to the International Primary CNS Lymphoma Collaborative Group (IPCG) efficacy assessment criteria.
Overall Survival (OS) | From the date of study enrollment until death from any cause, assessed up to 36 months.
  Overall Survival (OS):
  Defined as the time from study enrollment to death from any cause.
Cause of Death | From the date of study enrollment until death, categorized by cause, assessed up to 36 months.
  Disease-related Death: Includes death due to lymphoma or acute toxicity from treatment.
  Other Causes: Includes death due to cardiovascular disease, infections, accidents, second primary malignancies, undetermined mixed causes, or unknown causes.
Safety(Toxicity, AE, SAE)) | Monitored throughout the treatment period and until the end of the safety follow-up period, assessed up to approximately 12 months.
  Toxicity Reactions: Graded according to the NCI CTCAE (version 5.0) criteria, with the investigator determining whether the toxicity is treatment-related.
  Adverse Events (AE): Events that lead to an interruption of treatment for more than 3 days, or early termination of the study.
  Serious Adverse Events (SAE): Defined as per Section 5.1 of the protocol. Supportive Treatment: Any treatments administered to address toxicity reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Facility Name: The First Hospital of Jilin University, Changchun, China

IPD SHARING:
Plan to Share IPD: Undecided